CLINICAL TRIAL: NCT01748682
Title: Use of Very Low Calorie Liquid Diet in the Preoperative Phase of Bariatric Surgery
Brief Title: Very Low Calorie Liquid Diet for Pre op Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silvia Leite Faria (Other)
Collaborators: Gastrocirurgia, Brazil (Other); University of Brasilia (Other)
Responsible Party: Sponsor-Investigator, Silvia Leite Faria, Master in Human Nutrition, Gastrocirurgia, Brazil
Organization: Gastrocirurgia, Brazil (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Morbid Obesity; Steatosis
Keywords: Very low calorie diet; liquid diet; visceral fat; liver fat.
MeSH Terms: conditions — Obesity, Morbid; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquid Diet Group (Experimental): The group followed a very low calorie liquid diet for two weeks
  Interventions: Other: A very low calorie diet of two different consistencies
- Control Group (Active Comparator): The group followed a very low calorie diet of normal consistency for two weeks.
  Interventions: Other: A very low calorie diet of two different consistencies

INTERVENTIONS:
Other: A very low calorie diet of two different consistencies — Liquid and normal consistency diet with a very low calorie diet will be given to patients pre-operatively in bariatric surgery

SUMMARY:
Despite the relative consensus on the benefits of pre-surgical weight loss, i.e., the reduction of comorbidities associated with surgical act, such as decreased visceral fat, liver volume, hemorrhage perioperative and surgical time, the characteristics of the diet to be employed in this period need to be defined more clearly. As there is no description of comparative studies on diet of normal consistency, using solids and liquids, there are doubts as to the real need for consistency liquid diet in preoperative bariatric surgery. The lack of robust evidence has made nutrition professionals adopt different procedures. There is still a belief that these patients are unable to lose weight in the preoperative period, the ongoing history of previous attempts without success.

ELIGIBILITY:
Inclusion Criteria:

* To be clinically severe obese; To be in preoperative phase of bariatric surgery.

Exclusion Criteria:

* Pregnancy and minors under 18 and adults over 60 years of age.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Loss of body weight | 2 weeks
  The patients were weighed at the start and after following a liquid diet for tow weeks they were weighed again.

SECONDARY OUTCOMES:
Total body, visceral and liver fat loss, resting metabolic rate and changes in blood and urinary parameters | 2 weeks
  At the start, bioimpedance and indirect calorimetry exams, abdominal ultrasound scans, blood tests and urinary exams were made of the patients and after following a set diet for 2 weeks these measurements were taken again.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia L Faria, MSc, Principal Investigator — Gastrocirurgia of Brasilia
Locations (1):
- Gastrocirurgia de Brasilia, Brasília, Federal District, Brazil